CLINICAL TRIAL: NCT05630885
Title: A Limited-Center, Prospective, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Cenicriviroc Mesylate on Arterial Inflammation in People Living With HIV
Brief Title: A Study to Evaluate the Effects of Cenicriviroc Mesylate on Arterial Inflammation in People Living With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5415
Record Dates: First submitted 2022-11-10; First posted 2022-11-30 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: HIV-1-infection; Elevated Cardiovascular Risk
Keywords: HIV; Vascular Inflammation

STUDY DESIGN:
Intervention Model Description: At study entry, participants were randomized 2:1 to oral CVC (Arm A) or oral placebo for CVC (Arm B) once a day. The study treatment was added to the participants' pre-existing antiretroviral treatment (ART) regimens.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CVC arm (Arm A) (Experimental): Participants with pre-existing ART regimen of efavirenz (EFV) took CVC 300 mg. Participants with all other pre-existing ART regimens took CVC 150 mg.
  Interventions: Drug: CVC 150 mg; Drug: CVC 300 mg
- Placebo for CVC arm (Arm B) (Placebo Comparator): Participants with pre-existing ART regimen of efavirenz (EFV) took placebo for CVC 300 mg. Participants with all other pre-existing ART regimens took placebo for CVC 150 mg.
  Interventions: Other: Placebo for CVC 150 mg; Other: Placebo for CVC 300 mg

INTERVENTIONS:
Drug: CVC 150 mg — Administered as one 150-mg tablet by mouth once a day with food.
  Arms: CVC arm (Arm A)
Drug: CVC 300 mg — Administered as two 150-mg tablets by mouth once a day with food.
  Arms: CVC arm (Arm A)
Other: Placebo for CVC 150 mg — Administered as one 150-mg matching placebo tablets by mouth once a day with food.
  Arms: Placebo for CVC arm (Arm B)
Other: Placebo for CVC 300 mg — Administered as two 150-mg matching placebo tablets by mouth once a day with food.
  Arms: Placebo for CVC arm (Arm B)

SUMMARY:
The study was conducted to determine if cenicriviroc mesylate (CVC) would decrease vascular inflammation as measured by 18F-fluorodeoxyglucose (FDG)-positron emission tomography (PET)/computed tomography (CT) imaging of the aorta and carotid arteries.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled phase II clinical trial comparing the intervention of CVC versus placebo for a duration of 24 weeks on arterial inflammation evaluated by FDG-PET/CT imaging.

A total of 110 participants were randomized 2:1 to the CVC arm (Arm A) or placebo for CVC arm (Arm B). Stratification by statin use at randomization ensured even distribution of statin use between the treatment groups.

Analyses were based on the efficacy population: all enrolled participants who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.

Analysis of the primary outcome utilized multiple imputation by regression to impute missing data.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented to be living with HIV-1 infection.
2. Currently on a stable, continuous NNRTI-based or unboosted INSTI-based ART regimen for ≥48 weeks prior to study entry with no plans to change ART during the course of the study.
3. At least a year of controlled HIV-1 RNA levels.
4. Current CD4+ cell count >200 cells/mm^3.
5. Elevated cardiovascular risk defined as at least one of the following:

   * Clinical atherosclerotic disease (symptomatic atherosclerotic lesions in any vessel)
   * Subclinical atherosclerotic disease (coronary artery calcification [CAC] >10 or presence of non-obstructive plaques)
   * Diabetes mellitus (DM) or prediabetes
   * Obesity
   * Hypertension or blood pressure ≥130/80 mmHg
   * Elevated LDL cholesterol (fasting LDL of >160 mg/dL)
   * Low HDL cholesterol (<40 mg/dL)
   * Current tobacco smoking
   * Family history of premature coronary artery disease (CAD)
   * hsCRP >2.0 mg/L

Key Exclusion Criteria:

1. Acute coronary syndrome
2. A current diagnosis of latent or active tuberculosis (TB) infection
3. Current diagnosis with other intracellular pathogens (Mycobacterium avium complex, Listeria monocytogenes, Toxoplasma gondii, and Cryptococcus neoformans).
4. Untreated hepatitis B virus (HBV) infection
5. Current hepatitis C virus (HCV) infection
6. Current, acute or clinically significant infection or illness requiring IV antibiotics or hospitalization
7. History of cirrhosis with severe hepatic impairment and/or hepatic decompensation
8. Active malignancy, except squamous cell skin cancer.
9. Hemoglobin A1c >8% within 90 days prior to study entry.
10. Initiation of statin therapy or change in statin dose within 90 days prior to study entry.
11. Current use of any of the statins at the doses indicated:

    * Atorvastatin, >40 mg/day dose
    * Rosuvastatin, ≥20 mg/day dose
12. Concurrent use of drugs with potential drug-drug interactions with CVC within 90 days prior to study entry.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Lo, MD, MMSc, Study Chair — Massachusetts General Hospital
Locations (19):
- United States (19):
  - University of California, Los Angeles CARE Center CRS (Site # 601), Los Angeles, California
  - UCSD Antiviral Research Center CRS (Site # 701), San Diego, California
  - UCSF HIV/AIDS CRS (Site # 801), San Francisco, California
  - Harbor University of California Los Angeles Center CRS (Site # 603), Torrance, California
  - Northwestern University CRS (Site # 2701), Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS) (Site # 101), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics (BWH TCRS) CRS (Site # 107), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS (Site # 2101), St Louis, Missouri
  - Weill Cornell Chelsea CRS (Site # 7804), New York, New York
  - Weill Cornell Uptown CRS (Site # 7803), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (Site # 31787), Rochester, New York
  - Chapel Hill CRS (Site # 3201), Chapel Hill, North Carolina
  - Cincinnati CRS (Site # 2401), Cincinnati, Ohio
  - Case CRS (Site # 2501), Cleveland, Ohio
  - Ohio State University CRS (Site # 2301), Columbus, Ohio
  - University of Pittsburgh CRS (Site # 1001), Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS (Site # 3652), Nashville, Tennessee
  - Houston AIDS Research Team CRS (Site # 31473), Houston, Texas
  - University of Washington Positive Research CRS (Site # 1401), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NHLBI BioData Catalyst® (BDC) (including data dictionaries and case report forms).
Supporting Information: Study Protocol, SAP
Time Frame: Within 3 years of final participant follow-up.
Access Criteria: Data will be available by request in the NHLBI repository.
URL: https://biodatacatalyst.nhlbi.nih.gov/

REFERENCES:
- See also: Specific table used in the study protocol. For example, "The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009)." — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 participants were enrolled from 19 US clinical research sites between May 30, 2023 and January 5, 2024.
Pre-assignment Details: Participants were randomized 2:1 to CVC arm (Arm A) or placebo for CVC arm (Arm B) and stratified by statin use status (current statin use or no current statin use) at study entry (enrollment).
Groups:
- CVC Arm (Arm A): Participants with pre-existing ART regimen of EFV took CVC 300 mg. Participants with all other pre-existing ART regimens took CVC 150 mg.
  CVC 150 mg: Administered as one 150-mg tablet by mouth once a day with food.
  CVC 300 mg: Administered as two 150-mg tablets by mouth once a day with food.
- Placebo for CVC Arm (Arm B): Participants with pre-existing ART regimen of EFV took placebo for CVC 300 mg. Participants with all other pre-existing ART regimens took placebo for CVC 150 mg.
  Placebo for CVC 150 mg: Administered as one 150-mg matching placebo tablets by mouth once a day with food.
  Placebo for CVC 300 mg: Administered as two 150-mg matching placebo tablets by mouth once a day with food.
Period: Study Completion
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Started | 74 | 36
Completed (Participants who have been in the study for at least 22 weeks are considered to have completed the study.) | 70 | 36
Not Completed | 4 | 0
Not completed — Took prohibited medications | 2 | 0
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Efficacy Analysis Population Set
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Started (Efficacy population: all enrolled participants who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.) | 70 | 36
Completed | 59 | 34
Not Completed | 11 | 2
Not completed — Took prohibited medications | 3 | 1
Not completed — Prematurely discontinued study treatment before week 22 | 8 | 1

BASELINE CHARACTERISTICS:
Population: Population is based on enrolled participants who initiated study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B) | Total
Number analyzed (Participants) | 74 | 36 | 110
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [51 to 62] | 58 [54 to 65] | 58 [53 to 63]
Age, Customized [Count of Participants; unit: Participants]
  Age Groups: 45-54 | 25 | 11 | 36
  Age Groups: 55-64 | 37 | 16 | 53
  Age Groups: 65-74 | 12 | 8 | 20
  Age Groups: 75+ | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 7 | 30
  Male | 51 | 29 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 61 | 28 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 12 | 38
  White | 46 | 24 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Gender Identity [Count of Participants; unit: Participants]
  Cisgender | 72 | 36 | 108
  Transgender Spectrum | 2 | 0 | 2
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.5 [25.5 to 32.2] | 28.7 [24.6 to 33.2] | 28.5 [25.1 to 32.8]
BMI Groups [Count of Participants; unit: Participants]
  Underweight (< 18.5) | 0 | 0 | 0
  Normal (18.5 - 24.9) | 16 | 11 | 27
  Overweight (25 - 29.9) | 31 | 8 | 39
  Obese (30+) | 27 | 17 | 44
Estimated Glomerular Filtration Rate (eGFR) [Median (Inter-Quartile Range); unit: mL/min/1.73m^2] — Estimated glomerular filtration rate (eGFR) calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation.
  mL/min/1.73m^2 | 86 [73 to 95] | 77 [65 to 89] | 82 [70 to 94]
eGFR Groups [Count of Participants; unit: Participants] — Estimated glomerular filtration rate (eGFR) calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation.
  Participants
    < 60 | 3 | 3 | 6
    60 - < 90 | 39 | 25 | 64
    90+ | 32 | 8 | 40
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 656 [504 to 900] | 681 [539 to 794] | 666 [508 to 888]
CD4 Percent [Median (Inter-Quartile Range); unit: %] | 35.3 [30.0 to 45.0] | 34.0 [28.9 to 41.0] | 34.8 [30.0 to 43.6]
HIV-1 RNA [Count of Participants; unit: Participants] — HIV-1 RNA levels were quantified at Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory using an ultrasensitive viral load (VL) assay. Assays with lower limit of quantification (LLQ) of 20, 30, 40, and 50 copies/mL were reported.
  Participants
    < Lower Limit of Quantification (LLQ) | 70 | 31 | 101
    ≥ Lower Limit of Quantification (LLQ) | 4 | 5 | 9
Antiretroviral Therapy (ART) Class [Count of Participants; unit: Participants]
  INSTI-based | 53 | 27 | 80
  NNRTI-based | 12 | 7 | 19
  INSTI and NNRTI-based | 9 | 2 | 11
Count of High-Risk Cardiovascular Risk Factors [Count of Participants; unit: Participants]
  One | 12 | 4 | 16
  Two | 21 | 7 | 28
  Three | 18 | 10 | 28
  Four or more | 23 | 15 | 38
Statin-use at Entry [Count of Participants; unit: Participants]
  Current-use of Statins | 42 | 19 | 61
  No Current-use of Statins | 32 | 17 | 49
Index Vessel [Count of Participants; unit: Participants] — Index vessel is the most inflamed vessel (highest target vessel target-to-background ratio (TBR) between aorta, left, or right carotid) at study entry. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Participants
    number analyzed (Participants) | 58 | 32 | 90
    Aorta | 45 | 23 | 68
    Left Carotid Artery | 6 | 3 | 9
    Right Carotid Artery | 7 | 6 | 13
Index Vessel Most-Diseased Segment (MDS) Target-to-Background Ratio (TBR) [Median (Inter-Quartile Range); unit: Ratio] — Index vessel MDS TBR is the most-diseased (inflamed) segment of the index vessel. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Ratio
    number analyzed (Participants) | 58 | 32 | 90
    (all) | 2.26 [2.05 to 2.54] | 2.22 [1.93 to 2.42] | 2.23 [2.00 to 2.48]
Aorta Vessel TBR [Median (Inter-Quartile Range); unit: Ratio] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Ratio
    number analyzed (Participants) | 57 | 31 | 88
    (all) | 2.12 [1.90 to 2.40] | 2.02 [1.76 to 2.32] | 2.10 [1.82 to 2.34]
Left Carotid Artery Vessel TBR [Median (Inter-Quartile Range); unit: Ratio] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Ratio
    number analyzed (Participants) | 46 | 21 | 67
    (all) | 1.75 [1.65 to 1.94] | 1.80 [1.69 to 2.04] | 1.76 [1.67 to 2.00]
Right Carotid Artery Vessel TBR [Median (Inter-Quartile Range); unit: Ratio] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Ratio
    number analyzed (Participants) | 47 | 22 | 69
    (all) | 1.81 [1.64 to 1.90] | 1.82 [1.70 to 1.96] | 1.81 [1.66 to 1.91]
Bilateral Carotid Arteries Vessel TBR [Median (Inter-Quartile Range); unit: Ratio] — Obtained by averaging the right carotid and left carotid artery vessel TBR for a given participant. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Ratio
    number analyzed (Participants) | 46 | 21 | 67
    (all) | 1.78 [1.64 to 1.96] | 1.78 [1.72 to 2.03] | 1.78 [1.68 to 1.96]
Aorta Vessel Standard Uptake Value (SUV) [Median (Inter-Quartile Range); unit: SUV] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  SUV
    number analyzed (Participants) | 57 | 33 | 90
    (all) | 1.85 [1.68 to 2.25] | 1.94 [1.70 to 2.35] | 1.92 [1.68 to 2.29]
Bilateral Carotid Arteries Vessel SUV [Median (Inter-Quartile Range); unit: SUV] — Obtained by averaging the right carotid and left carotid artery vessel SUV for a given participant. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  SUV
    number analyzed (Participants) | 51 | 21 | 72
    (all) | 1.58 [1.41 to 1.92] | 1.79 [1.59 to 2.06] | 1.65 [1.45 to 1.97]
C-Reactive Protein (hsCRP) [Median (Inter-Quartile Range); unit: mg/L] — Measured using high-sensitivity CRP (hsCRP) test to detect smaller changes in CRP levels. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  mg/L
    number analyzed (Participants) | 58 | 33 | 91
    (all) | 1.44 [0.62 to 3.33] | 2.69 [1.15 to 6.08] | 1.71 [0.70 to 5.17]
Interleukin-6 [Median (Inter-Quartile Range); unit: pg/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  pg/mL
    number analyzed (Participants) | 58 | 33 | 91
    (all) | 1.57 [0.94 to 2.51] | 2.02 [1.38 to 3.02] | 1.79 [1.08 to 2.55]
Soluble CD14 [Median (Inter-Quartile Range); unit: ng/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  ng/mL
    number analyzed (Participants) | 58 | 33 | 91
    (all) | 1403 [1233 to 1703] | 1435 [1271 to 1779] | 1415 [1246 to 1729]
Soluble CD163 [Median (Inter-Quartile Range); unit: ng/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  ng/mL
    number analyzed (Participants) | 57 | 34 | 91
    (all) | 729 [556 to 938] | 720 [480 to 930] | 729 [498 to 938]
MCP-1 [Median (Inter-Quartile Range); unit: pg/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  pg/mL
    number analyzed (Participants) | 58 | 33 | 91
    (all) | 171 [140 to 206] | 184 [145 to 228] | 175 [140 to 209]
MIP-1 alpha [Count of Participants; unit: Participants] — Assay lower limit of quantification (LLQ) is 46.9 pg/mL. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Participants
    number analyzed (Participants) | 59 | 34 | 93
    < Lower Limit of Quantification (LLQ) | 58 | 33 | 91
    Missing | 1 | 1 | 2
MIP-1 beta [Count of Participants; unit: Participants] — Assay lower limit of quantification (LLQ) is 31.3 pg/mL. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  Participants
    number analyzed (Participants) | 59 | 34 | 93
    < Lower Limit of Quantification (LLQ) | 10 | 4 | 14
    ≥ Lower Limit of Quantification (LLQ) | 48 | 29 | 77
    Missing | 1 | 1 | 2
MIP-1 beta [Median (Inter-Quartile Range); unit: pg/mL] — Records below LLQ are imputed as half of LLQ. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  pg/mL
    number analyzed (Participants) | 58 | 33 | 91
    (all) | 52.1 [34.6 to 71.2] | 55.3 [36.6 to 64.2] | 52.4 [36.1 to 66.6]
RANTES [Median (Inter-Quartile Range); unit: ng/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  ng/mL
    number analyzed (Participants) | 57 | 34 | 91
    (all) | 69.7 [50.1 to 105] | 70.2 [50.6 to 94.4] | 69.7 [50.1 to 98.6]
Fasting Glucose [Median (Inter-Quartile Range); unit: mg/dL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  mg/dL
    number analyzed (Participants) | 59 | 34 | 93
    (all) | 95 [86 to 102] | 95 [89 to 108] | 95 [87 to 104]
Fasting Insulin [Median (Inter-Quartile Range); unit: uIU/mL] — Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  uIU/mL
    number analyzed (Participants) | 58 | 34 | 92
    (all) | 9.02 [5.01 to 15.9] | 10.4 [7.25 to 17.9] | 9.90 [6.30 to 16.0]
Homeostasis Model Assessment-estimated Insulin Resistance (HOMA-IR) [Median (Inter-Quartile Range); unit: HOMA-IR Index] — HOMA-IR is a calculation used to assess insulin resistance and is calculated with the formula: insulin (uIU/mL) * glucose (mg/dL) / 405. Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
  HOMA-IR Index
    number analyzed (Participants) | 53 | 32 | 85
    (all) | 2.01 [1.33 to 3.84] | 2.50 [1.55 to 4.89] | 2.35 [1.33 to 3.97]

OUTCOME MEASURES:

1. Primary Outcome: Change (Expressed as Ratio to Baseline) in 18-FDG-PET Target-to-background Ratio (TBR) of the Most Diseased Segment (MDS) of the Index (Most-inflamed) Vessel.
Description: Target-to-Background Ratio (TBR) measures the intensity of inflammation of a target arterial wall (aorta, left carotid, right carotid), relative to its respective blood background. Specifically, it is the ratio of the Standardized Uptake Value (SUV) of 18-FDG-PET in the target vessel to SUV in the blood background. A negative number for the change in TBR means a reduction in the target arterial wall inflammation over time.
  Index vessel is the vessel with the highest vessel TBR at baseline.
  The most diseased segment is the approximately 1-cm section of the vessel with the highest activity at baseline.
  The results are expressed as the ratio of TBR at week 24 to baseline.
  For the statistical analyses, results for the 6 and 9 missing values in Arm A and Arm B, respectively, were imputed using multiple imputation by regression.
Time Frame: Measured at baseline and week 24
Population: Efficacy population: all enrolled participants who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 53 | 25
Fold-change | 0.95 [0.85 to 1.01] | 0.93 [0.87 to 1.02]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the MDS of the index vessel, adjusting for statin-use. The study was powered to detect a between-group difference of 0.046 in log10 MDS TBR (10% relative fold-change), assuming a null difference of 0 in log10 MDS TBR (a ratio of 1 in absolute-scale), a standard deviation of 0.065 of change in log10 TBR, and 75 evaluable participants; Test type: Superiority; p = 0.65, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use. Analysis used multiple imputation for missing data; Slope = 0.984, 95% CI 2-sided [0.916 to 1.056] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale and rounded to 3 decimal places. It reflects the relative geometric mean fold-change in the TBR from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the MDS of the index vessel differently by statin-use at study entry (use versus no-use); Test type: Other — Statistical test for interaction; p = 0.40, Regression, Linear — P-value for modification of the CVC treatment effect by subgroups defined by statin-use is presented. A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use and its interaction with treatment. Analysis used multiple imputation for missing data
Statistical Analysis 3: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the MDS of the index vessel differently by sex (female versus male); Test type: Other — Statistical test for interaction; p = 0.63, Regression, Linear — P-value for modification of the CVC treatment effect by subgroups defined by sex is presented. A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for sex (F vs M) and its interaction with treatment. Analysis used multiple imputation for missing data
Statistical Analysis 4: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the MDS of the index vessel differently by race (Black/African-American versus Non-Black/African-American); Test type: Other — Statistical test for interaction; p = 0.71, Regression, Linear — P-value for modification of the CVC treatment effect by subgroups defined by race is presented. A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for race and its interaction with treatment. Analysis used multiple imputation for missing data

2. Secondary Outcome: Change (Expressed as Ratio to Baseline) in Aortic TBR (and Other TBRs)
Description: Target-to-Background Ratio (TBR) measures the intensity of inflammation of a target arterial wall (aorta, left carotid, right carotid), relative to its respective blood background. Specifically, it is the ratio of the Standard Uptake Value (SUV) of 18-FDG-PET in the target vessel to SUV in the blood background. A negative number for the change in TBR implies a reduction in the target arterial wall inflammation over time.
  The results are expressed as the ratio of TBR at week 24 to baseline.
Time Frame: Measured at baseline and week 24
Population: Efficacy population with evaluable records: all enrolled participants with evaluable records who completed at least 22 weeks of study treatment and remained on the same ART drug class throughout the study without use of prohibited medications.
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 55 | 27
Fold-change
  Aorta TBR: number analyzed (Participants) | 52 | 24
  Aorta TBR | 1.00 [0.93 to 1.09] | 0.99 [0.91 to 1.11]
  Bilateral Carotid TBR: number analyzed (Participants) | 40 | 16
  Bilateral Carotid TBR | 0.99 [0.89 to 1.09] | 1.02 [0.89 to 1.11]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the aorta adjusting for statin-use; Test type: Superiority; p = 0.91, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 0.996, 95% CI 2-sided [0.930 to 1.067] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the right and left carotid arteries adjusting for statin-use; Test type: Superiority; p = 0.64, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 0.980, 95% CI 2-sided [0.901 to 1.066] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change (Expressed as Ratio to Baseline) in Standardized Uptake Value (SUV) Measured in the Carotid Arteries and Aorta
Description: Standard Uptake Value (SUV) measures the intensity of inflammation of a target arterial wall (aorta, left carotid, right carotid). Specifically, it is the average of all evaluable SUV for a given arterial vessel. A negative number for the change in SUV implies a reduction in the target arterial wall inflammation over time.
  The results are expressed as the ratio of SUV at week 24 to baseline.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 56 | 28
Fold-change
  Aorta SUV: number analyzed (Participants) | 52 | 26
  Aorta SUV | 1.00 [0.93 to 1.11] | 1.00 [0.88 to 1.10]
  Bilateral Carotid SUV: number analyzed (Participants) | 49 | 18
  Bilateral Carotid SUV | 1.02 [0.94 to 1.11] | 1.00 [0.89 to 1.06]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes arterial inflammation in the aorta adjusting for statin-use; Test type: Superiority; p = 0.79, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.010, 95% CI 2-sided [0.939 to 1.087] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale and rounded to 3 decimal places. It reflects the relative geometric mean fold-change in the SUV from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.69, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.017, 95% CI 2-sided [0.935 to 1.106] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose (mg/dL) measures the level of sugar (glucose) in the blood after fasting (no eating or drinking except water) for at least 8 hours. Higher value of change means an increase in glucose levels over time.
  The results are expressed as the change in fasting glucose from baseline to week 24.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 58 | 34
mg/dL | 1.00 [-9.00 to 8.00] | -0.50 [-13.00 to 8.00]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of fasting glucose adjusting for statin-use; Test type: Superiority; p = 0.49, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Model adjusted for statin-use; Slope = 2.5, 95% CI 2-sided [-4.6 to 9.6] — Estimate reflects the relative mean change in fasting glucose from baseline for CVC compared to placebo

5. Secondary Outcome: Change (Expressed as Ratio to Baseline) in Fasting Insulin and Homeostasis Model Assessment-estimated Insulin Resistance (HOMA-IR)
Description: Insulin is a hormone crucial in regulating blood sugar levels. HOMA-IR is a calculation used to assess insulin resistance and is calculated with the formula: insulin (uIU/mL) * glucose (mg/dL) / 405. Higher value of change in insulin and HOMA-IR means an increase in insulin resistance over time.
  The results are expressed as the ratio of fasting insulin or HOMA-IR at week 24 to baseline.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 58 | 33
Fold-change
  Fasting insulin | 0.91 [0.67 to 1.28] | 0.89 [0.57 to 1.31]
  HOMA-IR: number analyzed (Participants) | 52 | 31
  HOMA-IR | 0.85 [0.63 to 1.37] | 0.90 [0.46 to 1.48]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of fasting insulin adjusting for statin-use; Test type: Superiority; p = 0.62, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.07, 95% CI 2-sided [0.81 to 1.43] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in fasting insulin from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of HOMA-IR adjusting for statin-use; Test type: Superiority; p = 0.61, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.09, 95% CI 2-sided [0.78 to 1.54] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in HOMA-IR from baseline for CVC compared to placebo

6. Secondary Outcome: Change (Expressed as Ratio to Baseline) in Biomarkers of Inflammation (IL-6, hsCRP, and MCP-1)
Description: The cytokine, Interleukin-6 (IL-6, pg/mL); protein, high-sensitivity C Reactive Protein (hsCRP, mg/L); and chemokine, monocyte chemoattractant protein-1 (MCP-1, pg/mL) are all markers of inflammation. Higher value of change means an increase in the biomarker levels over time. Higher levels of these biomarkers indicates inflammation.
  MCP-1 is a ligand of CCR2 that was expected to increase with CVC.
  The results are expressed as the ratio of hsCRP, IL-6, or MCP-1 at week 24 to baseline.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 58 | 33
Fold-change
  hsCRP | 0.85 [0.51 to 1.30] | 0.84 [0.61 to 1.48]
  Interleukin-6 | 0.99 [0.78 to 1.64] | 1.10 [0.71 to 1.56]
  MCP-1 | 5.00 [3.96 to 6.04] | 0.99 [0.86 to 1.36]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of hsCRP adjusting for statin-use; Test type: Superiority; p = 0.91, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 0.97, 95% CI 2-sided [0.62 to 1.52] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in hsCRP from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes the levels of IL-6 adjusted for statin-use; Test type: Superiority; p = 0.94, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.01, 95% CI 2-sided [0.77 to 1.33] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in IL-6 from baseline for CVC compared to placebo
Statistical Analysis 3: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes the levels of MCP-1 adjusting for statin-use; Test type: Superiority; p < 0.001, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 4.74, 95% CI 2-sided [3.89 to 5.77] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in MCP-1 from baseline for CVC compared to placebo

7. Secondary Outcome: Change in Biomarkers of Immune Activation (sCD14 and sCD163)
Description: The soluble proteins soluble-CD14 (sCD14, ng/mL) and soluble-CD163 (sCD163, ng/mL) are all markers of monocyte/macrophage activation. Higher value of change means an increase in the biomarker levels over time. Higher levels of sCD14 and sCD163 occur in response to inflammation and infection.
  The results are expressed as the difference between sCD14 or sCD163 from baseline to week 24.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 58 | 33
ng/mL
  Soluble CD14 | -16.2 [-147 to 112] | 6.66 [-115 to 155]
  Soluble CD163: number analyzed (Participants) | 57 | 33
  Soluble CD163 | -21.8 [-93.9 to 50.5] | 17.4 [-67.3 to 68.8]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of sCD14 adjusting for statin-use; Test type: Superiority; p = 0.38, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Model adjusted for statin-use; Slope = -49, 95% CI 2-sided [-158 to 60] — Estimate reflects the relative mean change in sCD14 from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes the levels of sCD163 adjusting for statin-use; Test type: Superiority; p = 0.88, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Model adjusted for statin-use; Slope = -6.3, 95% CI 2-sided [-87 to 75] — Estimate reflects the relative mean change in sCD163 from baseline for CVC compared to placebo

8. Secondary Outcome: Change (Expressed as Ratio to Baseline) in Plasma Levels of Chemokine Receptor 5 (CCR5) Ligands (RANTES and MIP-1 Beta)
Description: The chemokines macrophage inflammatory protein-1 alpha and beta (MIP-1 alpha and beta, pg/mL) as well as the chemokine, RANTES (ng/mL), are markers of inflammation. Higher value of change means an increase in the biomarker levels over time. Higher levels of these biomarkers indicates inflammation.
  RANTES and MIP-1 beta are ligands of CCR5 that were expected to increase with CVC.
  The results are expressed as the ratio of RANTES or MIP-1 beta at week 24 to baseline.
Time Frame: Measured at baseline and week 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
Number analyzed (Participants) | 58 | 33
Fold-change
  MIP-1 beta | 2.44 [1.82 to 3.54] | 1.07 [0.92 to 2.07]
  RANTES: number analyzed (Participants) | 57 | 33
  RANTES | 0.98 [0.80 to 1.22] | 1.06 [0.92 to 1.29]
Statistical Analysis 1: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes the levels of MIP-1 beta adjusting for statin-use; Test type: Superiority; p < 0.001, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.65, 95% CI 2-sided [1.28 to 2.12] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in MIP-1 beta from baseline for CVC compared to placebo
Statistical Analysis 2: Comparison: CVC Arm (Arm A) vs Placebo for CVC Arm (Arm B); Evaluates whether CVC, compared to placebo, changes levels of RANTES adjusting for statin-use; Test type: Superiority; p = 0.85, Regression, Linear — A-priori threshold for statistical significance is at p < 0.05. No adjustments for multiple comparisons were done; Outcome was log10-transformed. Model adjusted for statin-use; Slope = 1.02, 95% CI 2-sided [0.82 to 1.28] — Estimate obtained from regression on log10-transformed scale was back-transformed to the original scale. It reflects the relative geometric mean fold-change in RANTES from baseline for CVC compared to placebo

ADVERSE EVENTS:
Time Frame: From study entry to completion at Week 24 or premature study discontinuation.
Description: All adverse events (AE) that met reporting criteria as defined in Protocol v2.0 Section 7.2 were collected. The DAIDS AE Grading Table (v2.1) was used. All eligible participants who initiated study treatment are included.
Arm/Group | CVC Arm (Arm A) | Placebo for CVC Arm (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/36
Serious Adverse Events (participants affected / at risk) | 4/74 | 2/36
Other Adverse Events (participants affected / at risk) | 44/74 | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVC Arm (Arm A) (N=74) | Placebo for CVC Arm (Arm B) (N=36)
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVC Arm (Arm A) (N=74) | Placebo for CVC Arm (Arm B) (N=36)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 6 | 2
Influenza (Infections and infestations) | 2 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 4 | 1
Blood cholesterol increased (Investigations) | 2 | 1
Blood creatinine decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 4 | 3
Blood sodium increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 2
Creatinine renal clearance decreased (Investigations) | 5 | 4
Glomerular filtration rate decreased (Investigations) | 21 | 5
Haemoglobin decreased (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form: Protocol Version 2.0 (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05630885/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT05630885/SAP_001.pdf